CLINICAL TRIAL: NCT04783753
Title: A Non-Randomized, Open-Label, Three-Part, Drug-Drug Interaction Study to Evaluate the Effects of Itraconazole, Carbamazepine, and Quinidine on the Pharmacokinetics and Safety of EDP-514 in Healthy Subjects
Brief Title: Drug-Drug Interaction Study Between EDP-514, Itraconazole, Carbamazepine, and Quinidine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 514-003
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B
Keywords: drug-drug interaction
MeSH Terms: conditions — Hepatitis B | interventions — Itraconazole; Carbamazepine; Quinidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EDP-514 and Itraconazole interaction (Part 1) (Experimental)
  Interventions: Drug: EDP-514; Drug: Itraconazole
- EDP-514 and Carbamazepine interaction (Part 2) (Experimental)
  Interventions: Drug: EDP-514; Drug: Carbamazepin
- EDP-514 and Quinidine interaction (Part 3) (Experimental)
  Interventions: Drug: EDP-514; Drug: Quinidine

INTERVENTIONS:
Drug: EDP-514 — Subjects will receive EDP-514 on Days 1 and 14
  Arms: EDP-514 and Itraconazole interaction (Part 1)
Drug: EDP-514 — Subjects will receive EDP-514 on Days 1 and 23
  Arms: EDP-514 and Carbamazepine interaction (Part 2)
Drug: EDP-514 — Subjects will receive EDP-514 on Days 1 and 8
  Arms: EDP-514 and Quinidine interaction (Part 3)
Drug: Itraconazole — Subjects will receive itraconazole QD for 14 days
  Arms: EDP-514 and Itraconazole interaction (Part 1)
Drug: Carbamazepin — Subjects will receive carbamazepine BID for 23 days
  Arms: EDP-514 and Carbamazepine interaction (Part 2)
Drug: Quinidine — Subjects will receive quinidine BID for 8 days
  Arms: EDP-514 and Quinidine interaction (Part 3)

SUMMARY:
Non-randomized, 3-part, open-label, drug-drug interaction (DDI) study to evaluate the effect of itraconazole, carbamazepine, or quinidine on the PK and safety of EDP-514 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive
* Female subjects who are heterosexually active and of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 30 days after the last dose of EDP-514.
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of clinically significant active infection.
* A positive urine drug screen at Screening or Day -1.
* Current tobacco smokers or use of tobacco products within 3 months prior to Screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).

  • Clinically significant laboratory abnormalities at screening or Day -1, as determined by the Investigator (including but not limited to hypokalemia, hypocalcemia, or hypomagnesemia for Part 3 participants).
* History of regular alcohol consumption
* Participation in a clinical trial within 30 days prior to the first dose of study drug.

For Part 2 (Carbamazepine) participants:

* Participants of Asian ancestry, given association of carbamazepine and severe rash (Stevens Johnson Syndrome [SJS] and Toxic Epidermal Necrolysis [TEN]) with HLA-B 1502 in this population.
* Platelets, white blood cell count or hemoglobin below the lower limit of normal, due to reported incidence of agranulocytosis and aplastic anemia with carbamazepine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-514 with and without coadministration with itraconazole | up to 19 days
AUC of EDP-514 with and without coadministration with itraconazole | 19 days
Cmax of EDP-514 with and without coadministration with carbamazepine | up to 28 days
AUC of EDP-514 with and without coadministration with carbamazepine | up to 28 days
Cmax of EDP-514 with and without coadministration with quinidine | up to 13 days
AUC of EDP-514 with and without coadministration with quinidine | up to 13 days

SECONDARY OUTCOMES:
Safety measured by adverse events | up to 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Pharmaceutical Research Association, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No